CLINICAL TRIAL: NCT02553083
Title: High Dose Dual Therapy (HDDT) for Eradication of Helicobacter Pylori Infection
Acronym: HDDT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Yaron Niv, Chief of Gastroenterology, Deputy CEO RMC, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0380-15-RMC
Record Dates: First submitted 2015-07-26; First posted 2015-09-17 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Bacterial Infection Due to Helicobacter Pylori (H. Pylori)
MeSH Terms: interventions — Esomeprazole; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Nexium 40 mg and amoxicillin 1.5 gr twice daily for 14 days
  Interventions: Drug: Nexium 40 mg; Drug: amoxicillin 1.5 gr
- Group 2 (Active Comparator): Nexium 40 mg and doxycycline 200 mg twice daily for 14 days
  Interventions: Drug: Nexium 40 mg; Drug: doxycycline 200 mg
- Group 3 (Active Comparator): Nexium 20 mg, clarythromicin 500 mg, and amoxicillin 1 gr twice daily for 14 days
  Interventions: Drug: Nexium 20 mg; Drug: clarythromicin 500 mg; Drug: amoxicillin 1gr

INTERVENTIONS:
Drug: Nexium 40 mg — Nexium 40 mg twice daily for 14 days
  Arms: Group 1; Group 2
Drug: amoxicillin 1.5 gr — amoxicillin 1.5 gr twice daily for 14 days
  Arms: Group 1
Drug: doxycycline 200 mg — doxycycline 200 mg twice daily for 14 days
  Arms: Group 2
Drug: Nexium 20 mg — Nexium 20 mg twice a day for 10 days
  Arms: Group 3
Drug: clarythromicin 500 mg — clarythromicin 500 mg twice a day for 10 days
  Arms: Group 3
Drug: amoxicillin 1gr — amoxicillin 1gr twice a day for 10 days
  Arms: Group 3

SUMMARY:
The investigators will performed a large-scale multi center trial to compare the efficacy of a high-dose dual therapy (HDDT) with that of standard therapies in treatment-naive (n = 300) patients with Hp infection. Consecutive symptomatic patients will be recruited in Israel and Spain when tested positive to Hp with serology and 13C urea breath test (13C-UBT) due to symptoms. Patients with gastric cancer, MALT lymphoma, and younger than 18 or older than 80 years old will be excluded. All patients will be naive to eradication therapy and will be randomized into one of three groups:

Group 1: Nexium 40 mg and amoxicillin 1.5 gr twice daily for 14 days Group 2: Nexium 40 mg and doxycycline 200 mg twice a day Group 3: Triple therapy of Nexium 20 mg, clarythromycin 500 mg, and amoxicillin 1gr twice a day for 10 days (regular accepted treatment).

All treatments will be stopped for a month and then 13CUBT will be repeated. The primary aim of the study is to assess eradication success, intentioned to treat and per protocol in the three treatment regimens.

The secondary aim of the study is to assess the safety of high dose amoxicillin and doxycycline.

DETAILED DESCRIPTION:
Introduction High dose dual therapy (HDDT) for Helicobacter pylori (Hp) eradication was successfully tried in Taiwan for naive as well as experienced patients who failed a previous trial. This new approach relies on the rare resistance of Hp to amoxicillin which is about 1% all over the world. High intra gastric pH increases the efficacy of amoxicillin, thus the "old" dual therapy with a proton pump inhibitor and amoxicillin, but now in high doses for a longer time, has a potential to achieve a high eradication rate. Yang and co investigators randomized 450 naïve and 168 treatment-experienced patients in Taiwan, all infected by Hp, for HDDT, sequential and triple therapies. In the intention-to-treat analysis, Hp was eradicated in 95.3%, 85.3% and 80.7%, respectively in naïve, and 89.3%, 51.8% and 78.6%, respectively in experienced patients. No more adverse events were found in the HDDT group. They divided the high dose of amoxicillin into 4 doses a day. This approach may be unnecessary since Kim and colleagues demonstrated the same results when the same dose of amoxicillin was divided into 2 or 4 times a day. Recently doxcycylin was found effective in triple or quadruple therapy regimens with no adverse effect in the high dose of 200 mg BID.

The investigators will try that approach, successful in Asian patients, in a collaborative study that included Spanish and Israeli patients. The investigators will investigate whether a combination of a high-dose proton pump inhibitor and amoxicillin (dual therapy) will be more effective than standard first-line 10 days triple therapy in eradicating Hp. Since patients who are allergic to penicillin cannot be treated with amoxicillin The investigators will compare HDDT amoxicillin-based therapy also with HDDT doxycycline -based therapy.

Protocol

The investigators will performed a large-scale multi center trial to compare the efficacy of a high-dose dual therapy (HDDT) with that of standard therapies in treatment-naive (n = 300) patients with Hp infection. Consecutive symptomatic patients will be recruited in Israel and Spain when tested positive to Hp with serology and 13CUBT due to symptoms. Patients with gastric cancer, MALT lymphoma, and younger than 18 or older than 80 years old will be excluded. All patients will be naive to eradication therapy and will be randomized into one of three groups:

Group 1: Nexium 40 mg and amoxicillin 1.5 gr twice daily for 14 days Group 2: Nexium 40 mg and doxycycline 200 mg twice a day Group 3: Triple therapy of Nexium 20 mg, clarythromycin 500 mg, and amoxicillin 1gr twice a day for 10 days (regular accepted treatment).

All treatments will be stopped for a month and then 13CUBT will be repeated. The primary aim of the study is to assess eradication success, intentioned to treat and per protocol in the three treatment regimens.

The secondary aim of the study is to assess the safety of high dose amoxicillin and doxycycline .

Hypothesis The investigators hypothesize that the success rate of eradication therapy in groups 1 and 2 will be significantly better than of group 3, with a good safety profile. If so, HDDT will be the answer for Hp eradication in areas with high Clarithromycin and metronidazole resistance.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected with Helicobacter pylori

Exclusion Criteria:

* Patients with gastric cancer or MALT lymphoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-10-22 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | 2 weeks therapy
  Eradication rate

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Niv, MD, Principal Investigator — RMC
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel